CLINICAL TRIAL: NCT00333151
Title: Effect on Glycemic Control of Liraglutide in Combination With Rosiglitazone Plus Metformin Versus Rosiglitazone Plus Metformin in Subjects With Type 2 Diabetes
Brief Title: Effect of Liraglutide on Blood Glucose Control in Subjects With Type 2 Diabetes
Acronym: LEAD-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1574
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Rosiglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: liraglutide
Drug: rosiglitazone
Drug: metformin

SUMMARY:
This trial is conducted in the United States of America (USA) and Canada. This trial is designed to show the effect of treatment with liraglutide when added to existing rosiglitazone and metformin combination therapy and to compare it with the effects of therapy with rosiglitazone and metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Treated with oral anti-diabetic (OAD) drugs for at least 3 months
* Treated with one or more OAD and in moderate to poor glycemic control
* Body Mass Index (BMI) less than or equal to 45.0 kg/m2

Exclusion Criteria:

* Treatment with insulin within the last three months prior to the trial except due to intercurrent illness, at the discretion of the Investigator
* Any serious medical condition
* Treatment with any drug that could interfere with glucose level

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 26 weeks of treatment

SECONDARY OUTCOMES:
body weight
Safety and tolerability
Glycaemic control

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (79):
- United States (62):
  - Novo Nordisk Investigational Site, Goodyear, Arizona
  - Novo Nordisk Investigational Site, Colton, California
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Mission Viejo, California
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Santa Ana, California
  - Novo Nordisk Investigational Site, Santa Barbara, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, New Britain, Connecticut
  - Novo Nordisk Investigational Site, Washington D.C., District of Columbia
  - Novo Nordisk Investigational Site, Fort Myers, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Lake Mary, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Athens, Georgia
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Powder Springs, Georgia
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, New Albany, Indiana
  - Novo Nordisk Investigational Site, Des Moines, Iowa
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Baton Rouge, Louisiana
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Tupelo, Mississippi
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Reno, Nevada
  - Novo Nordisk Investigational Site, Berlin, New Jersey
  - Novo Nordisk Investigational Site, Plainsboro, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Brooklyn, New York
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, Rochester, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Durham, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Kettering, Ohio
  - Novo Nordisk Investigational Site, Mentor, Ohio
  - Novo Nordisk Investigational Site, Duncan, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Lubbock, Texas
  - Novo Nordisk Investigational Site, Midland, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Canada (17):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Ottawa, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Laval, Quebec
  - Novo Nordisk Investigational Site, Gatineau
  - Novo Nordisk Investigational Site, Mississauga
  - Novo Nordisk Investigational Site, Montreal
  - Novo Nordisk Investigational Site, Québec
  - Novo Nordisk Investigational Site, Red Deer
  - Novo Nordisk Investigational Site, St. John's
  - Novo Nordisk Investigational Site, Toronto
  - Novo Nordisk Investigational Site, Vancouver
  - Novo Nordisk Investigational Site, Windsor

REFERENCES:
- [Background] Buse JB, Garber A, Rosenstock J, Schmidt WE, Brett JH, Videbaek N, Holst J, Nauck M. Liraglutide treatment is associated with a low frequency and magnitude of antibody formation with no apparent impact on glycemic response or increased frequency of adverse events: results from the Liraglutide Effect and Action in Diabetes (LEAD) trials. J Clin Endocrinol Metab. 2011 Jun;96(6):1695-702. doi: 10.1210/jc.2010-2822. Epub 2011 Mar 30. PMID 21450987
- [Result] Sullivan SD, Alfonso-Cristancho R, Conner C, Hammer M, Blonde L. Long-term outcomes in patients with type 2 diabetes receiving glimepiride combined with liraglutide or rosiglitazone. Cardiovasc Diabetol. 2009 Feb 26;8:12. doi: 10.1186/1475-2840-8-12. PMID 19245711
- [Result] Zinman B, Gerich J, Buse JB, Lewin A, Schwartz S, Raskin P, Hale PM, Zdravkovic M, Blonde L; LEAD-4 Study Investigators. Efficacy and safety of the human glucagon-like peptide-1 analog liraglutide in combination with metformin and thiazolidinedione in patients with type 2 diabetes (LEAD-4 Met+TZD). Diabetes Care. 2009 Jul;32(7):1224-30. doi: 10.2337/dc08-2124. Epub 2009 Mar 16. PMID 19289857
- [Result] McGill JB. Insights from the Liraglutide Clinical Development Program--the Liraglutide Effect and Action in Diabetes (LEAD) studies. Postgrad Med. 2009 May;121(3):16-25. doi: 10.3810/pgm.2009.05.1998. PMID 19491536
- [Result] Blonde L, Russell-Jones D. The safety and efficacy of liraglutide with or without oral antidiabetic drug therapy in type 2 diabetes: an overview of the LEAD 1-5 studies. Diabetes Obes Metab. 2009 Dec;11 Suppl 3:26-34. doi: 10.1111/j.1463-1326.2009.01075.x. PMID 19878259
- [Result] Bode BW, Brett J, Falahati A, Pratley RE. Comparison of the efficacy and tolerability profile of liraglutide, a once-daily human GLP-1 analog, in patients with type 2 diabetes >/=65 and <65 years of age: a pooled analysis from phase III studies. Am J Geriatr Pharmacother. 2011 Dec;9(6):423-33. doi: 10.1016/j.amjopharm.2011.09.007. Epub 2011 Nov 4. PMID 22055210
- [Result] Henry RR, Buse JB, Sesti G, Davies MJ, Jensen KH, Brett J, Pratley RE. Efficacy of antihyperglycemic therapies and the influence of baseline hemoglobin A(1C): a meta-analysis of the liraglutide development program. Endocr Pract. 2011 Nov-Dec;17(6):906-13. doi: 10.4158/ep.17.6.906. PMID 22193143
- [Result] Zinman B, Schmidt WE, Moses A, Lund N, Gough S. Achieving a clinically relevant composite outcome of an HbA1c of <7% without weight gain or hypoglycaemia in type 2 diabetes: a meta-analysis of the liraglutide clinical trial programme. Diabetes Obes Metab. 2012 Jan;14(1):77-82. doi: 10.1111/j.1463-1326.2011.01493.x. Epub 2011 Oct 30. PMID 21883806
- [Result] Niswender K, Pi-Sunyer X, Buse J, Jensen KH, Toft AD, Russell-Jones D, Zinman B. Weight change with liraglutide and comparator therapies: an analysis of seven phase 3 trials from the liraglutide diabetes development programme. Diabetes Obes Metab. 2013 Jan;15(1):42-54. doi: 10.1111/j.1463-1326.2012.01673.x. Epub 2012 Sep 9. PMID 22862847
- [Result] Alves C, Batel-Marques F, Macedo AF. A meta-analysis of serious adverse events reported with exenatide and liraglutide: acute pancreatitis and cancer. Diabetes Res Clin Pract. 2012 Nov;98(2):271-84. doi: 10.1016/j.diabres.2012.09.008. Epub 2012 Sep 23. PMID 23010561
- [Result] King AB, Montanya E, Pratley RE, Blonde L, Svendsen CB, Donsmark M, Sesti G. Liraglutide achieves A1C targets more often than sitagliptin or exenatide when added to metformin in patients with type 2 diabetes and a baseline A1C <8.0%. Endocr Pract. 2013 Jan-Feb;19(1):64-72. doi: 10.4158/EP12232.OR. PMID 23186975
- [Result] Jensen TM, Saha K, Steinberg WM. Is there a link between liraglutide and pancreatitis? A post hoc review of pooled and patient-level data from completed liraglutide type 2 diabetes clinical trials. Diabetes Care. 2015 Jun;38(6):1058-66. doi: 10.2337/dc13-1210. Epub 2014 Dec 12. PMID 25504028
- [Result] Davidson JA, Orsted DD, Campos C. Efficacy and safety of liraglutide, a once-daily human glucagon-like peptide-1 analogue, in Latino/Hispanic patients with type 2 diabetes: post hoc analysis of data from four phase III trials. Diabetes Obes Metab. 2016 Jul;18(7):725-8. doi: 10.1111/dom.12653. Epub 2016 Apr 28. PMID 26936426
- [Derived] Fonseca VA, Devries JH, Henry RR, Donsmark M, Thomsen HF, Plutzky J. Reductions in systolic blood pressure with liraglutide in patients with type 2 diabetes: insights from a patient-level pooled analysis of six randomized clinical trials. J Diabetes Complications. 2014 May-Jun;28(3):399-405. doi: 10.1016/j.jdiacomp.2014.01.009. Epub 2014 Jan 21. PMID 24561125
- [Derived] Hegedus L, Moses AC, Zdravkovic M, Le Thi T, Daniels GH. GLP-1 and calcitonin concentration in humans: lack of evidence of calcitonin release from sequential screening in over 5000 subjects with type 2 diabetes or nondiabetic obese subjects treated with the human GLP-1 analog, liraglutide. J Clin Endocrinol Metab. 2011 Mar;96(3):853-60. doi: 10.1210/jc.2010-2318. Epub 2011 Jan 5. PMID 21209033
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com